# Statistical Analysis Plan (SAP) Official Title:

# Comparison of Complication Rates of Onlay vs Sublay Mesh Repair of Incisional Hernia Brief Title:

Complication Rate of Onlay vs Sublay Mesh Repair in Incisional Hernia

#### ClinicalTrials.gov Identifier:

NCT ID: Not Yet Assigned

#### **Organization's Unique Protocol ID:**

HMC-QAD-F No. IREB-1221

#### **Study Type:**

Interventional Study (Randomized Controlled Trial)

#### **Study Design:**

Parallel Assignment, Open Label

#### **Sponsor:**

Hayatabad Medical Complex, Peshawar, Pakistan

#### **Responsible Party:**

Principal Investigator

#### **Principal Investigator:**

Dr. Gohar Ali Principal Investigator Department of Surgery Hayatabad Medical Complex, Peshawar, Pakistan

#### **Planned Statistical Analysis:**

Comparative analysis of postoperative complication rates between onlay and sublay mesh repair techniques using appropriate descriptive and inferential statistical methods.

#### **Ethics Approval:**

Approved by Ethical Committee, Hayatabad Medical Complex, Peshawar

Approval Number: HMC-QAD-F No. IREB-1221

# **Analysis Population:**

- All randomized patients
- Per-protocol population for sensitivity analysis

## **Descriptive Statistics:**

- Continuous variables: mean  $\pm$  SD or median (IQR)
- Categorical variables: frequency (%)

## **Primary Outcome Analysis:**

- Compare **postoperative complication rate** between onlay and sublay groups
- Statistical Test: Chi-square or Fisher's exact test
- Significance level:  $\alpha = 0.05$

# **Secondary Outcome Analysis:**

- 1. Hernia recurrence: Chi-square test; Kaplan-Meier curves for time-to-recurrence
- 2. Length of hospital stay: Independent t-test or Mann-Whitney U test
- 3. Operative time: Independent t-test or Mann-Whitney U test

# **Subgroup Analysis (optional):**

- Stratified by age group ( $40 \text{ vs} \ge 40$ )
- Stratified by BMI (<30 vs 30–40)

# **Handling Missing Data:**

- Multiple imputation if missing >5%
- Sensitivity analysis comparing complete case vs imputed dataset

#### **Software:**

• Analysis performed using SPSS version 23

# **Reporting:**

- Two-sided p-values
- 95% confidence intervals for effect estimates
- Tables and figures for primary and secondary outcomes